CLINICAL TRIAL: NCT00417339
Title: A Multicentric Observational Trial on Protein Bound Uremic Toxins in Nocturnal Hemodialysis
Brief Title: Protein-bound Uremic Retention Solutes and Long Nocturnal Hemodialysis: a Longitudinal Analysis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Björn Meijers, Prof, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: NHD002
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: End Stage Kidney Disease
Keywords: hemodialysis; dialysis adequacy; uremic retention solute
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine, dialysate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- hemodialysis, 4h, twice weekly: hemodialysis, four hours, twice weekly
  Interventions: Procedure: hemodialysis
- hemodialysis, 8h, twice weekly: hemodialysis, eight hours, twice weekly
  Interventions: Procedure: hemodialysis
- hemodialysis, 8h, every other day: hemodialysis, eight hours, every other day
  Interventions: Procedure: hemodialysis
- hemodialysis, 8h, six days per week: hemodialysis, eight hours, six days per week
  Interventions: Procedure: hemodialysis

INTERVENTIONS:
Procedure: hemodialysis — individualised

SUMMARY:
Study on intradialytic kinetics of protein-bound uremic retention solutes during long nocturnal hemodialysis

DETAILED DESCRIPTION:
Although remarkable progress has been made, chronic kidney disease still poses a major burden on both individual patients, as well as on society as a whole. There is a strong inverse relationship between decreasing renal function, as estimated by glomerular filtration rate, and mortality rate, especially death due to cardiovascular disease. The exact cause(s) remain to be elucidated. Uremic toxins might play an important role.

In the course of decreasing renal function the concentration of numerous intracellular and extracellular compounds vary from the non-uremic state. A still increasing number of uremic retention solutes are being identified. Renal replacement strategies aim to remove potentially harmful substances from the body. Traditionally much attention has been paid to small water-soluble molecules such as urea nitrogen and creatinine. Based on the results of the recent HEMO and ADEMEX studies, increases of small water-soluble solute removal above the level reached with modern dialysis techniques (HD, PD) seem not to be advantageous with regard to patient outcome. These findings may point to the importance of other distinct groups of uremic retention solutes. In view of the data described above, protein-bound solutes might be good candidates.

Several advantages of long duration hemodialysis have been observed, including a better control of blood pressure by decreasing extracellular fluid volume, lowering peripheral vascular resistance and improving endothelium-dependent and -independent vasodilation. A normalization of heart rate variability and improvement of left-ventricular function was noted as well. Furthermore, anemia control has been shown to be easier and several nutritional parameters improved in patients treated with long duration HD. The therapy results in higher small water-soluble solute removal, phosphate removal and greater elimination of larger molecules (e.g. β2-microglobulin).

It seems an appealing question whether a better control of the serum levels of protein-bound solutes can be achieved by long duration (nocturnal) hemodialysis. This might be another advantage of this therapeutic modality, or may even in part explain the better outcome of patients treated this way.

The study compares intermittent hemodialysis with long nocturnal hemodialysis with respect to serum concentrations of several protein bound uremic toxins, as well as solute removal.

ELIGIBILITY:
Inclusion Criteria:

* Start hemodialysis during 2007
* Age over 18 years
* Informed consent

Exclusion Criteria:

* Non consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: maintenance dialysis patients
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2006-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Björn KI Meijers, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Pieter Evenepoel, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven; Tom Dejagere, MD, Principal Investigator — Virga Jesse Ziekenhuis; Nigel Toussaint, MD, Principal Investigator — Geelong Hospital
Locations (4):
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Geelong Hospital, Geelong, Victoria
- Belgium (2):
  - Universitaire Ziekenhuizen Leuven, Leuven, Brabant
  - Virga Jesseziekenhuis, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bammens B, Evenepoel P, Keuleers H, Verbeke K, Vanrenterghem Y. Free serum concentrations of the protein-bound retention solute p-cresol predict mortality in hemodialysis patients. Kidney Int. 2006 Mar;69(6):1081-7. doi: 10.1038/sj.ki.5000115. PMID 16421516
- [Background] Fagugli RM, De Smet R, Buoncristiani U, Lameire N, Vanholder R. Behavior of non-protein-bound and protein-bound uremic solutes during daily hemodialysis. Am J Kidney Dis. 2002 Aug;40(2):339-47. doi: 10.1053/ajkd.2002.34518. PMID 12148107
- [Background] Pierratos A. Daily nocturnal home hemodialysis. Kidney Int. 2004 May;65(5):1975-86. doi: 10.1111/j.1523-1755.2004.00603.x. No abstract available. PMID 15086951